CLINICAL TRIAL: NCT03442569
Title: Phase II Multicenter Trial of Panitumumab, Nivolumab, and Ipilimumab for KRAS/NRAS/BRAF Wild-type MSS Refractory Metastatic Colorectal Adenocarcinoma
Brief Title: PhII Trial Panitumumab, Nivolumab, Ipilimumab in Kras/Nras/BRAF Wild-type MSS Refractory mCRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1632
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Panitumumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: This will be a single-arm, open-label, multicenter Phase II clinical trial investigating the clinical efficacy of nivolumab, ipilimumab, and panitumumab in subjects with unresectable refractory KRAS/NRAS/BRAF wild-type microsatellite stable metastatic colorectal cancer after an initial safety lead-in cohort to ensure the three drug combination is well-tolerated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label, single arm, Phase II (Experimental): Nivolumab and ipilimumab with panitumumab
  Interventions: Drug: Panitumumab; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Panitumumab — 6 mg/kg via IV every 2 weeks in combination with nivolumab and ipilimumab
  Other Names: Vectibix
Drug: Nivolumab — 240 mg via IV every 2 weeks in combination with panitumumab and ipilimumab
  Other Names: Opdivo
Drug: Ipilimumab — 1 mg/kg via IV every 6 weeks in combination with nivolumab and panitumumab
  Other Names: Yervoy

SUMMARY:
To investigate the combination of nivolumab and ipilimumab with panitumumab in subjects with unresectable, refractory, KRAS/NRAS/BRAF wild-type, microsatellite stable (MSS) metastatic colorectal cancer.

DETAILED DESCRIPTION:
The investigators will conduct a single-arm, open-label Phase II clinical trial investigating the combination of nivolumab and ipilimumab with panitumumab in subjects with unresectable, refractory, KRAS/NRAS/BRAF wild-type, microsatellite stable (MSS) metastatic colorectal cancer (mCRC). There will be an initial safety lead-in cohort to ensure the combination is well-tolerated. The primary objective of this study is to estimate the overall response rate in these subjects at 12 weeks . Secondary objectives include the following: estimating the overall response rate in these subjects at 12 weeks by immune-related RECIST criteria (irRECIST), estimating the best response rate by both RECIST 1.1 and irRECIST criteria, estimating progression-free survival (PFS) and duration of response using both RECIST 1.1 and irRECIST criteria, estimating overall survival (OS), and characterizing the safety issues associated with this regimen. Exploratory objectives involve investigating various biomarkers and peripheral blood and tumor assays.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed colorectal adenocarcinoma, with unresectable metastatic or locally advanced disease documented on diagnostic imaging studies.
2. Previously received 1-2 prior lines of therapy. Subjects who relapse within 6 months of adjuvant chemotherapy comprised of oxaliplatin and a fluoropyrimidine will have their adjuvant therapy count as one prior line of therapy.
3. Confirmed wild-type in KRAS and NRAS codons 12, 13, 59, 61, 117, and 146; and BRAF codon 600, by standard of care testing of tumor specimen. Tissue used for testing may have been collected from primary or metastatic site.
4. Microsatellite stable as detected by PCR-based assay or CLIA-certified sequencing methodology such as Foundation One; or mismatch repair proficient as detected by immunohistochemistry showing intact nuclear staining of MLH1, MSH2, MSH6, and PMS2
5. Radiographically measurable disease present per RECIST 1.1
6. Age ≥ 18 years at the time of consent.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
8. Blood counts performed within 3 weeks prior to starting study therapy must have absolute neutrophil count ≥ 1,500/mm3, platelets ≥ 100,000/mm3, and hemoglobin ≥ 9 g/dL.

   *Note: Hematology and other lab parameters that are ≤ grade 2 but still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.
9. Liver function tests performed within 3 weeks prior to starting study therapy must have total bilirubin ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase and aspartate aminotransferase ≤ 3 x ULN, and albumin ≥ 2.5 g/dL.
10. Serum creatinine performed within 3 weeks prior to starting study therapy must be ≤ 1.5 x ULN, or have calculated creatinine clearance (using Cockcroft-Gault formula provided in Appendix 11.3) of ≥ 50 mL/minute.
11. Females of childbearing potential must have a negative serum pregnancy test within 24 hours prior to receiving the first dose of study medication. Females of childbearing potential must agree to use 2 methods of effective contraception or abstain from heterosexual sex throughout the treatment period and for 5 months after the last dose of study treatment. Females of childbearing potential are women who have not been surgically sterilized (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or have not been free of menses for >1 year.
12. Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 7 months after the last dose of study treatment.
13. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
14. An adequate amount of archival tumor tissue must be available at baseline to be eligible for enrollment in the study. If archival tissue is not available or is inadequate, then the subject must consent to undergo a mandatory biopsy at baseline in order to participate in the study.

Exclusion Criteria:

1. Past treatment with an antibody targeting EGFR including cetuximab or panitumumab.
2. Past treatment with an antibody targeting immune checkpoints including CTLA-4, PD-1, PD-L1, PD-L2, or CD137.
3. Known untreated brain metastasis or brain metastasis treated within 3 months prior to enrollment in this trial.
4. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
5. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease free for at least five years.
6. Treatment within 21 days of the first dose of study drug with any other chemotherapy, immunotherapy, biologic therapy, vaccine therapy, or investigational treatment for the treatment of malignancy, or failure to recover from adverse effects of prior therapies administered over 4 weeks prior to Study Day 1. All toxicities from prior therapies must be ≤ Grade 1 (or ≤ Grade 2 for alopecia or peripheral neuropathy). Prior systemic treatment in the adjuvant setting is allowed. See note above under inclusion 3.1.8
7. Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent, or compliance to the study procedures.
8. Pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment. (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
9. History of organ allograft or other history of immunodeficiency, or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of investigational treatment.
10. Inability or unwillingness to comply with study and/or follow-up requirements.
11. Any major surgery, extensive radiotherapy, chemotherapy with clinically significant delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to randomization and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to randomization.
12. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug.
13. Known Human Immunodeficiency Virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV) infection. Subjects with laboratory evidence of cleared HBV and HCV infection will be permitted.
14. Active autoimmune disease requiring systemic treatment in the past 3 months (for example with disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators, local steroid injections, or inhaled or topical steroids would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
15. Active infection requiring intravenous systemic therapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna K Sanoff, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 medical institutions between March 2018 and June 2020.
Pre-assignment Details: A total of 61 subjects were consented to the trial, but 5 were deemed to be ineligible during screening and therefore were not enrolled on the trial.
Period: Overall Study
Arm/Group | Open-label, Single Arm, Phase II
Started | 56
Started Treatment | 55
Completed | 55
Not Completed | 1
Not completed — Subject was ineligible after enrollment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 56
Age, Customized [Count of Participants; unit: Participants]
  Age: 30-39 | 1
  Age: 40-49 | 9
  Age: 50-59 | 25
  Age: 60-69 | 17
  Age: 70-79 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 44
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) = CR + PR Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: 12 weeks
Population: Seven participants were unevaluable for the primary endpoint at 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 49
percentage of participants | 32 [21 to 45]

2. Secondary Outcome: Overall Response Rate Per irRECIST
Description: Overall Response Rate (ORR) = irCR + irPR Per immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) for target and/or non-target lesions and assessed by imaging: Complete Response (irCR), Disappearance of all lesions, no new lesions, lymph nodes < 10 mm in short axis; Partial Response (irPR), ≥30% decrease in the sum of target lesions and non-target lesions are irNN; Stable response (irSD), not meeting criteria for irCR, irPR, or irPD; Progressive Disease (irPD), ≥20% increase in tumor burden and minimum 5 mm absolute increase in compared to nadir; for no new non-target or (irNN) and where irPR or irPD are confirmed by a repeat, consecutive assessment no less than 4 weeks later
Time Frame: 12 weeks
Population: Seven participants were unevaluable for the primary endpoint at 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 49
percentage of participants | 34 [23 to 47]

3. Secondary Outcome: Median Progression Free Survival
Description: Median Progression Free Survival is the time at which 50% of the study population has experienced disease progression as defined by RECIST, irRECIST, or death from any cause.
Time Frame: Up to 3 years
Population: Participants initiated the study and were assessed for disease progression or survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 49
months | 6 [5.5 to 7.4]

4. Secondary Outcome: Median Overall Survival
Description: Time from the first day of treatment until death from any cause.
Time Frame: Up to 3 years
Population: Participants initiated the study and were assessed for survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 49
months | 17.4 [14.2 to 27.5]

5. Secondary Outcome: Median Duration of Response
Description: Duration of response is the time from documentation of tumor response to disease progression.
Time Frame: Up to 3 years
Population: Participants initiated the study and were assessed for response and disease progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 56
months | 5 [3.3 to 9]

6. Secondary Outcome: Toxicity of Treatment
Description: The number of treatment-emergent grade 3 and 4 toxicities as defined by the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03) was reported.
Time Frame: Up to 36 month
Population: Participants started to study the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label, Single Arm, Phase II
Number analyzed (Participants) | 56
Participants
  Blood and lymphatic system disorders - Other, specify | 3
  Hemolysis | 1
  Myocarditis | 1
  Adrenal insufficiency | 3
  Endocrine disorders - Other, specify | 1
  Abdominal pain | 2
  Colitis | 1
  Colonic obstruction | 1
  Constipation | 1
  Diarrhea | 3
  Gastrointestinal disorders - Other, specify | 2
  Nausea | 3
  Pancreatitis | 1
  Rectal pain | 1
  Small intestinal obstruction | 1
  Vomiting | 3
  Fatigue | 2
  Cholecystitis | 1
  Allergic reaction | 1
  Autoimmune disorder | 1
  Infections and infestations - Other, specify | 2
  Papulopustular rash | 1
  Paronychia | 1
  Rash pustular | 1
  Sepsis | 2
  Soft tissue infection | 1
  Alanine aminotransferase increased | 3
  Aspartate aminotransferase increased | 3
  Lipase increased | 5
  Lymphocyte count decreased | 4
  Neutrophil count decreased | 1
  Platelet count decreased | 1
  Serum amylase increased | 4
  White blood cell decreased | 2
  Anorexia | 1
  Dehydration | 1
  Hyperglycemia | 1
  Hypocalcemia | 2
  Hypokalemia | 4
  Hypomagnesemia | 8
  Hyponatremia | 1
  Hypophosphatemia | 4
  Pain in extremity | 1
  Headache | 1
  Delirium | 2
  Psychiatric disorders - Other, specify | 1
  Acute kidney injury | 1
  Urinary retention | 1
  Dyspnea | 2
  Hypoxia | 1
  Pneumonitis | 1
  Rash acneiform | 6
  Rash maculo-papular | 3
  Skin and subcutaneous tissue disorders - Other, specify | 1
  Stevens-Johnson syndrome | 1
  Surgical and medical procedures - Other, specify | 1
  Hypertension | 6
  Hypotension | 1
  Thromboembolic event | 2

ADVERSE EVENTS:
Time Frame: From Day 1 of treatment up to 3 years after completion of treatment
Arm/Group | Open-label, Single Arm, Phase II
All-Cause Mortality (participants affected / at risk) | 27/56
Serious Adverse Events (participants affected / at risk) | 21/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Single Arm, Phase II (N=56)
Abdominal pain (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Fatigue (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Myocarditis (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Sepsis (Infections and infestations) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
pancreatitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Single Arm, Phase II (N=56)
Abdominal pain (Gastrointestinal disorders) | 9
Acute kidney injury (Renal and urinary disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 3
Akathisia (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 17
Alkaline phosphatase increased (Investigations) | 15
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Anal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 16
Anorexia (Metabolism and nutrition disorders) | 19
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 20
Autoimmune disorder (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 6
Blurred vision (Eye disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Chills (General disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Conjunctivitis (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Creatinine increased (Investigations) | 1
Cushingoid (Endocrine disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 18
Dizziness (Nervous system disorders) | 6
Dry eye (Eye disorders) | 3
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 17
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Edema limbs (General disorders) | 6
Endocrine disorders - Other, specify (Endocrine disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Esophageal infection (Infections and infestations) | 1
Esophagitis (Gastrointestinal disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Eye pain (Eye disorders) | 1
Eyelid function disorder (Eye disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 24
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 16
Flatulence (Gastrointestinal disorders) | 1
Floaters (Eye disorders) | 1
Flu like symptoms (General disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Gastroparesis (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 10
Hematuria (Renal and urinary disorders) | 3
Hemoglobin increased (Investigations) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 21
Hyperthyroidism (Endocrine disorders) | 7
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 20
Hypomagnesemia (Metabolism and nutrition disorders) | 38
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 12
Hypotension (Vascular disorders) | 3
Hypothyroidism (Endocrine disorders) | 15
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
INR increased (Investigations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 7
Infusion related reaction (General disorders) | 4
Insomnia (Psychiatric disorders) | 5
Investigations - Other, specify (Investigations) | 8
Lethargy (Nervous system disorders) | 1
Lipase increased (Investigations) | 10
Lymphocyte count decreased (Investigations) | 21
Malaise (General disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Middle ear inflammation (Ear and labyrinth disorders) | 1
Mucosal infection (Infections and infestations) | 2
Mucositis oral (Gastrointestinal disorders) | 13
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nail infection (Infections and infestations) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 21
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 7
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 11
Penile pain (Reproductive system and breast disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 11
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Presyncope (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 27
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 51
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Rash pustular (Infections and infestations) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 3
Rectal pain (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Scleral disorder (Eye disorders) | 1
Serum amylase increased (Investigations) | 8
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 12
Skin infection (Infections and infestations) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Thromboembolic event (Vascular disorders) | 3
Upper respiratory infection (Infections and infestations) | 2
Urinary frequency (Renal and urinary disorders) | 4
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 21
Watering eyes (Eye disorders) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03442569/Prot_SAP_000.pdf